CLINICAL TRIAL: NCT07331584
Title: Effects of Elastic Band Versus Free Weight Resistance Training on Functional Capacity, Pulmonary Functioning and Quality of Life in Phase 2 of CABG Patients.
Brief Title: Elastic Band Versus Free Weight Resistance Training in Phase 2 of CABG Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fatima Shoaib
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: CABG
Keywords: coronary artery bypass graft, resistance training, functional residual capacities, pulmonary function test, quality of life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dumbell (Experimental): Group A will receive the exercises from dumb bells we will focus on both upper limb and lower limb the total session would be of 20-30 minutes, will be focusing on chest (pectoralis major), back (latissimus dorsi, rhomboids), legs (quadriceps, hamstring, glutes) and core (abdominals, lower back) and after that 5-7 min of cool down. Dyspnea will be measured.
  Interventions: Other: dumbell; Other: thera band
- elastic band (Experimental): Group B will receive the exercise form elastic band (TheraBand) for both upper limb and lower limb. Total session time would be 30 minutes will be focusing on chest (pectoralis major), back (latissimus dorsi, rhomboids), legs (quadriceps, hamstring, glutes) and core (abdominals, lower back) 10-12 reps and 1 set in starting progressively increased to 3 reps after that at the end of session 5-7 min cool down and gentle stretching 2 times per week for 12 weeks. Dyspnea should be monitored.
  Interventions: Other: dumbell; Other: thera band

INTERVENTIONS:
Other: dumbell — Group A will receive the exercises from dumb bells we will focus on both upper limb and lower limb the total session would be of 20-30 minutes, will be focusing on chest (pectoralis major), back (latissimus dorsi, rhomboids), legs (quadriceps, hamstring, glutes) and core (abdominals, lower back) and after that 5-7 min of cool down. Dyspnea will be measured.
Other: thera band — Group B will receive the exercise form elastic band (TheraBand) for both upper limb and lower limb. Total session time would be 30 minutes will be focusing on chest (pectoralis major), back (latissimus dorsi, rhomboids), legs (quadriceps, hamstring, glutes) and core (abdominals, lower back) 10-12 reps and 1 set in starting progressively increased to 3 reps after that at the end of session 5-7 min cool down and gentle stretching 2 times per week for 12 weeks. Dyspnea should be monitored.

SUMMARY:
The aim of this study compares the effects of elastic band and free weights on functional capacity, lung function and quality of life in phase 2 coronary artery bypass grafting patients. Resistance training is vital in cardiac rehabilitation for improving physical function, strength, and independence. These patients typically experience reduced functional capacity and lung function due to post-surgical deconditioning and inactivity, which can also impact quality of life.Determining whether elastic bands or free weights provide greater benefits in these areas may help optimize cardiac rehabilitation protocols by identifying a safe, effective, and accessible approach for improving patient outcomes. This research has the potential to guide evidence-based resistance training in post- coronary artery bypass grafting rehabilitation, ultimately supporting recovery and enhancing quality of life of patients.

DETAILED DESCRIPTION:
Patients who undergo cardiac surgery frequently faces pulmonary complications. This study aims to compare the effects of elastic band and free weights on functional capacity, lung function and quality of life in phase 2 coronary artery bypass grafting patients. Resistance training is vital in cardiac rehabilitation for improving physical function, strength, and independence. These patients typically experience reduced functional capacity and lung function due to post-surgical deconditioning and inactivity, which can also impact quality of life. Determining whether elastic bands or free weights provide greater benefits in these areas may help optimize cardiac rehabilitation protocols by identifying a safe, effective, and accessible approach for improving patient outcomes.

This research has the potential to guide evidence-based resistance training in post- coronary artery bypass grafting rehabilitation, ultimately supporting recovery and enhancing quality of life of patients. By comparing the effects of elastic band versus free weights resistance training on functional capacity, pulmonary functioning and quality of life in phase 2 of coronary artery bypass grafting. It will be a randomized clinical trial. Age of selected patients will be between 45 to 65 years and data will be collected from them. There will be two groups i.e. group A will receive 10 min walk warm up after that resistance training of upper and lower limb by using dumb bells and group B will receive 10 min of walk as warm up after that resistance training of upper and lower limb by using elastic band. International physical activity questionnaire used for quality of life, 6 min walk test for functional capacity and forced expiratory volume, forced vital capacity and peak expiratory flow rate for lung functioning.

Trial will be completed in 12 weeks (2x/week) after patients got discharged 4-8 weeks after the surgery and before and after each session, primary and secondary outcomes will be measured for both groups. After data collection, data will be analyzed using SPSS version 25

ELIGIBILITY:
Inclusion Criteria:

Male and female

* Age (45-64)
* Stable cardio vascular status
* Able to participate in mild to moderate exercise
* Must be in 4-8 week of CABG and medically cleared for phase 2.
* Able to provide informed consent

Exclusion Criteria:

Unstable cardiovascular condition.

* Pulmonary conditions
* Cognitive impairment
* Other major surgeries and comorbidities

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 Second | 12 weeks
  Forced Expiratory Volume in 1 Second (FEV1) is a key lung function test measuring how much air you can forcefully blow out in the first second of a deep breath, indicating how quickly your airways empty.
international physical activity questionnaire : Quality of life | 12 week
  The international physical activity questionnaire is a widely used tool designed to assess physical activity levels among adults. It evaluates various types of activity, including walking, moderateintensity activities, and vigorous-intensity activities, over the past week. The International Physical Activity Questionnaire (IPAQ) scoring involves converting reported activity (walking, moderate, vigorous) into MET-minutes per week by multiplying minutes by MET values (3.3 for walking, 4 for moderate, 8 for vigorous). Scores are then categorized as Low, Moderate, or High, based on specific criteria like achieving ≥3000 MET-min/week (High) or meeting minimum days/minutes for moderate activity (e.g., ≥3 days vigorous or ≥5 days moderate/walking for Moderate), to assess overall activity levels.
6 Minute Walk Test | 12 weeks
  A 6 min walk test is easier, safer to administer, better tolerated and better reflects activity of daily Living than another walk test. The 6-Minute Walk Test (6MWT) scoring primarily focuses on the total distance walked (6MWD) in meters, calculated by counting laps and adding any partial lap, noting rest times. Scores are interpreted using age/sex/height/weight-specific prediction equations (like those from the American Thoracic Society) to compare actual distance to expected normal, with lower scores indicating poorer function, though the longest distance from multiple tests is used to account for learning effects.
Forced Vital Capacity | 12 week
  FVC, or Forced Vital Capacity, is a key measurement in spirometry (lung function tests) that quantifies the total amount of air you can forcefully exhale from your lungs after taking the deepest breath
Peak Expiratory Flow Rate | 12 Week
  Peak Expiratory Flow Rate (PEFR) measures the fastest speed you can forcefully exhale air from your lungs

CONTACTS AND LOCATIONS:
Overall Officials: Riffat Malik, Principal Investigator — Riphah International University
Locations (1):
- Sehat Medical Complex Hanjerwal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No